CLINICAL TRIAL: NCT01989598
Title: A Phase 2 Study of Sequential Trametinib and GSK2141795 in Relapsed or Refractory Multiple Myeloma
Brief Title: Trametinib and Akt Inhibitor GSK2141795 in Treating Patients With Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-02148; NCI-2013-02148 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PHL-091; 9460 (Other: University Health Network-Princess Margaret Hospital); 9460 (Other: CTEP); N01CM00032 (NIH); UM1CA186644 (NIH); NCT01951495 (obsolete NCT alias)
Record Dates: First submitted 2013-11-18; First posted 2013-11-21 (Estimated); Results first posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Recurrent Plasma Cell Myeloma; Refractory Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — trametinib; GSK2141795

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (trametinib, Akt inhibitor GSK2141795) (Experimental): Patients receive trametinib orally PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients with progressive disease or who achieve less than PR after 4 courses may also receive Akt inhibitor GSK2141795 PO daily on days 1-28.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Trametinib; Drug: Uprosertib

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Drug: Trametinib — Given PO
  Other Names: GSK1120212; JTP-74057; MEK Inhibitor GSK1120212; Mekinist
Drug: Uprosertib — Given PO
  Other Names: GSK2141795; Oral Akt Inhibitor GSK2141795

SUMMARY:
This phase II trial studies how well trametinib and Akt inhibitor GSK2141795 work in treating patients with multiple myeloma that has come back (relapsed) or that does not respond to treatment (refractory). Trametinib and Akt inhibitor GSK2141795 may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the antitumor activity of trametinib determined by overall response rate (ORR) in patients that are stratified into groups based on: biomarker positive (neuroblastoma RAS viral [v-ras] oncogene homolog [NRAS], v-Ki-ras2 Kirsten rat sarcoma viral oncogene homolog [KRAS], v-raf murine sarcoma viral oncogene homolog B1 [BRAF] mutated) and biomarker negative (without NRAS, KRAS, BRAF mutation).

SECONDARY OBJECTIVES:

I. To evaluate progression free survival (PFS) and duration of response (DOR) in the two stratified groups.

II. To document ORR after the addition of GSK2141795 (Akt inhibitor GSK2141795) to trametinib in patients who have developed progressive disease or have achieved less than a partial response (PR) after 4 cycles of treatment.

III. To evaluate PFS and DOR in patients receiving trametinib plus GSK2141795. IV. To evaluate the safety profile of trametinib with and without GSK2141795.

TERTIARY OBJECTIVES:

I. To explore the relationship between clinical response and pharmacodynamic (PD) markers.

II. To explore the relationship between v-maf avian musculoaponeurotic fibrosarcoma oncogene homolog (MAF) expression as determined by quantitative polymerase chain reaction (qPCR), chromosomal abnormalities detected by florescence in situ hybridization (FISH), and clinical response.

III. To explore the role of integrin beta7 as a biomarker of MAF expression. IV. To explore the relationship between objective clinical response as well as progressive disease and the tumor mutational profile.

V. To explore mechanism of phosphatidylinositol 3 kinase (PI3K)/v-akt Murine Thymoma Viral Oncogene Homolog 1 (AKT) and retrovirus-associated deoxyribonucleic acid (DNA) sequence (RAS)-mitogen-activated protein kinase kinase (MEK)-mitogen-activated protein kinase 1 (ERK) activation and correlate these with clinical response and PD markers.

IV. To explore the feasibility of extracting circulating free tumor DNA (cfDNA) from peripheral blood and detecting RAS and RAF mutations using cfDNA.

OUTLINE:

Patients receive trametinib orally (PO) once daily (QD) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients with progressive disease or who achieve less than PR after 4 courses may also receive Akt inhibitor GSK2141795 PO daily on days 1-28.

After completion of study treatment, patients are followed up for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed multiple myeloma not otherwise specified (NOS) (10028566)
* Patients must have measurable disease as defined as at least one of the following (these baseline laboratory studies for determining eligibility must be obtained within 28 days prior to enrollment):

  * Serum M-protein >= 0.5 g/dl (>= 5 g/l)
  * Urine M-protein >= 200 mg/24 h
  * Serum free light chains (FLC) assay: involved FLC level >= 10 mg/dl (>= 100 mg/l) and an abnormal serum free light chain ratio (< 0.26 or > 1.65)
  * Biopsy proven plasmacytoma (should be measured within 28 days of first study drug administration); prior biopsy is acceptable
  * If the serum protein electrophoresis is unreliable for routine M-protein measurement, quantitative immunoglobulin levels on nephelometry or turbidimetry will be followed
* A diagnosis of multiple myeloma (MM) and documentation of relapsed or relapse/refractory status following at least 2 prior lines of therapy
* Documented laboratory (lab) results confirming tumor mutational status must be obtained at screening; patients in whom mutational status cannot be determined will be deemed ineligible
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Life expectancy of greater than 6 months
* Able to swallow and retain orally-administered medication and does not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels
* All prior treatment-related toxicities must be Common Terminology Criteria for Adverse Events (CTCAE) version (v)4 grade =< 1 (except alopecia) at the time of registration; subjects with toxicities attributed to prior anti-cancer therapy which are not expected to resolve and result in long lasting sequelae are permitted to enroll
* Absolute neutrophil count (ANC) >= 1.0 x 10^9/L
* Hemoglobin >= 8 g/dL
* Platelets >= 50 x 10^9/L
* Albumin >= 2.5 g/dL
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) (isolated bilirubin > 1.5 x ULN is acceptable if bilirubin is fractionated and direct bilirubin < 35%)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x institutional ULN
* Serum creatinine =< 1.5 mg/dL OR calculated creatinine clearance (Cockroft-Gault formula) >= 30 mL/min OR 24-hour urine creatinine clearance >= 30 mL/min
* Prothrombin time (PT)/international normalized ratio (INR) and partial thromboplastin time (PTT) =< 1.5 x institutional ULN
* Fasting serum glucose < 126 mg/dl (7 mmol/l)
* Left ventricular ejection fraction (LVEF) >= institutional lower limit of normal (LLN) by echocardiogram (ECHO) or multi gated acquisition scan (MUGA)
* Subjects that have been previously diagnosed with type 2 diabetes or steroid-induced diabetes must also meet the additional following criteria:

  * Diagnosed with diabetes >= 6 months prior to enrollment
  * Hemoglobin A1C (HbA1C) =< 8% at screening visit
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; women of child-bearing potential must have a negative serum pregnancy test within 7 days prior to the start of protocol therapy; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of trametinib administration
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* History of another malignancy; exception: patients who have been disease-free for 3 years, or patients with a history of completely resected non-melanoma skin cancer and/or patients with indolent second malignancies, are eligible; consult the Cancer Therapy Evaluation Program (CTEP) medical monitor if unsure whether second malignancies meet the requirements specified above
* History of interstitial lung disease or pneumonitis
* Diabetes mellitus currently requiring insulin; subjects with a history of steroid-induced hyperglycemia may be enrolled provided that HbA1C at screening visit is =< 8%
* Any major surgery, extensive radiotherapy, chemotherapy with delayed toxicity, biologic therapy, or immunotherapy within 28 days prior to randomization and/or daily or weekly chemotherapy or other approved anti-myeloma therapy without the potential for delayed toxicity within 14 days prior to registration
* Use of other investigational drugs within 28 days preceding the first dose of trametinib and during the study
* Symptomatic or untreated leptomeningeal or brain metastases or spinal cord compression
* Have a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to trametinib or excipients or to dimethyl sulfoxide (DMSO) or GSK214795
* Current use of a prohibited medication; the following medications or non-drug therapies are prohibited:

  * Other anti-cancer therapy while on study treatment; (note: megestrol [Megace] if used as an appetite stimulant is allowed)
  * Concurrent treatment with bisphosphonates is permitted; however, treatment must be initiated prior to the first dose of study therapy; prophylactic use of bisphosphonates in patients without bone disease is not permitted, except for the treatment of osteoporosis
  * The concurrent use of all herbal supplements is prohibited during the study (including, but not limited to, St. John's wort, kava, ephedra [ma huang], gingko biloba, dehydroepiandrosterone [DHEA], yohimbe, saw palmetto, or ginseng)
* In vitro data indicate that GSK2141795 is a cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) substrate; drugs that potently inhibit CYP3A4 could lead to increased GSK2141795 exposure in subjects, and should either be prohibited or used with caution; drugs which are strong inducers of cytochrome P450, family 3, subfamily A (CYP3A) and may result in lower exposures of GSK2141795 should also be prohibited; GSK2141795 also appears to be a moderate in vitro inhibitor of cytochrome P450, family 2, subfamily C, polypeptide 8 (CYP2C8) (50% inhibitory concentration [IC50] 3 mcM) and CYP3A4 (IC50 11 mcM); drugs that are substrates of CYP3A4 or CYP2C8 with a narrow therapeutic index may be prohibited; drugs that are sensitive substrates of CYP3A4 or CYP2C8 should be used with caution
* History or current evidence/risk of retinal vein occlusion (RVO) or retinal pigment epithelial detachment (RPED):

  * History of RVO or RPED, or predisposing factors to RVO or RPED (e.g., uncontrolled glaucoma or ocular hypertension, uncontrolled systemic disease such as hypertension, diabetes mellitus, or history of hyperviscosity or hypercoagulability syndromes)
  * Visible retinal pathology as assessed by ophthalmic exam that is considered a risk factor for RVO or RPED such as evidence of new optic disc cupping, evidence of new visual field defects, and intraocular pressure > 21 mmHg
* History or evidence of cardiovascular risk including any of the following:

  * Left ventricular ejection fraction (LVEF) < LLN
  * A QT interval corrected for heart rate using the Bazett's formula Fridericia corrected QT interval (QTcB) >= 480 msec (>= 500 msec for subjects with bundle branch block)
  * History or evidence of current clinically significant uncontrolled arrhythmias (exception: patients with controlled atrial fibrillation for > 30 days prior to randomization are eligible)
  * Other clinically significant electrocardiogram (ECG) abnormalities including second (2nd) degree (type II) or third (3rd) degree atrioventricular (AV) block
  * Subject with intra-cardiac defibrillators or pacemakers
  * History of acute coronary syndromes (including myocardial infarction and unstable angina), coronary angioplasty, or stenting within 6 months prior to randomization
  * History or evidence of current >= class II congestive heart failure as defined by the New York Heart Association (NYHA) functional classification system
  * Treatment-refractory hypertension defined as a blood pressure of systolic > 140 mmHg and/or diastolic > 90 mmHg which cannot be controlled by anti-hypertensive therapy
  * Known cardiac metastases
* Known human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV) infection (with the exception of chronic or cleared HBV and HCV infection, which will be allowed)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* The study drug must not be administered to pregnant women or nursing mothers; women of childbearing potential should be advised to avoid pregnancy and use effective methods of contraception; men with a female partner of childbearing potential must have either had a prior vasectomy or agree to use effective contraception; if a female patient or a female partner of a patient becomes pregnant while the patient receives trametinib, the potential hazard to the fetus should be explained to the patient and partner (as applicable); these potential risks may also apply to GSK2141795

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-10-30 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2020-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Trudel, Principal Investigator — University Health Network-Princess Margaret Hospital
Locations (5):
- Canada (5):
  - Foothills Hospital, Calgary, Alberta
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Kingston Health Sciences Centre, Kingston, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Trametinib, Akt Inhibitor GSK2141795): Patients receive trametinib orally PO QD (once daily) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients with progressive disease or who achieve less than PR after 4 courses may also receive Akt inhibitor GSK2141795 PO daily on days 1-28.
  Laboratory Biomarker Analysis: Correlative studies
  Pharmacological Study: Correlative studies
  Trametinib: Given PO
  Uprosertib: Given PO
Period: Overall Study
Arm/Group | Treatment (Trametinib, Akt Inhibitor GSK2141795)
Started | 25 (Includes pts receiving Single agent Trametinib and pts who are receiving Trametinib with AKT Inhibitor GSK2141795)
Dual Therapy With Trametinib and GSK2141795 | 12 (Patients with progressive disease or who achieve less than PR after 4 courses also received Akt inhibitor GSK2141795 PO daily on days 1-28 along with Tremetinib)
Completed | 25 (Note: 25 patients enrolled, however, one patient unevaluable was not included in analysis)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Trametinib, Akt Inhibitor GSK2141795)
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 12
Age, Continuous [Median (Full Range); unit: years] | 64 [42 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 25

OUTCOME MEASURES:

1. Primary Outcome: ORR Evidenced by Confirmed Response Rate, Defined as Number of Patients With Partial Response or Better by International Myeloma Working Group (IMWG) Criteria Divided by the Number of Patients in the Applicable Group (Biomarker Positive or Negative)
Description: "Per International Myeloma Working Group (IMWG) Criteria: Complete Response (CR), Negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and < 5% plasma cells in bone marrow; Partial Response (PR), > 50% reduction of serum M-protein and reduction in 24 hours urinary M-protein by >90% or to < 200 mg/24 h; Overall Response (OR) = CR + PR."
Time Frame: Every 4 weeks until progression or death, whichever occurs first, an average of 9 months.
Measure: Number; unit: participants
Groups:
- Treatment (Trametinib): Patients receive trametinib orally PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Treatment (Trametinib, Akt Inhibitor GSK2141795): Patients who develop progressive disease on trametinib monotherapy or achieve less then a PR after 4 cycles of treatment will have the option to continue on trametinib with the addition of GSK2141795
Arm/Group | Treatment (Trametinib) | Treatment (Trametinib, Akt Inhibitor GSK2141795)
Number analyzed (Participants) | 24 | 11
participants | 1 | 2

2. Secondary Outcome: PFS
Description: Summarized for each cohort using the Kaplan-Meier method, from the date of start of treatment to the date of documented progression (based on IMWG criteria) or death due to any cause, assessed every 4 weeks
Time Frame: Time from the date of start of treatment to the date of documented progression (based on IMWG criteria) or death, whichever occurs first, due to any cause, assessed every 4 weeks, an average of 9 months.
Population: Note: 25 patients enrolled, however, one patient unevaluable was not included in analysis
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Trametinib, Akt Inhibitor GSK2141795)
Number analyzed (Participants) | 24
months | 1.8 [0.9 to 3.2]

3. Secondary Outcome: DOR (Duration of Response)
Description: Summarized for each cohort using the Kaplan-Meier method.
Time Frame: From time measurement criteria are met for CR or PR (complete or partial response), (whichever recorded first) until first date that recurrent or progressive disease is objectively documented or to death due to multiple myeloma, assessed every 4 weeks
Population: Not reported. Data were not collected and not analyzed for this outcome measure.
Arm/Group | Treatment (Trametinib) | Treatment (Trametinib, Akt Inhibitor GSK2141795)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: ORR After the Addition of AKT Inhibitor GSK2141795 to Trametinib in Patients Who Have Developed Progressive Disease or Have Achieved Less Than a PR
Description: as for outcome 1
Time Frame: Every 4 weeks until progression or death, whichever occurs first, an average of 9 months.
Population: Trametinib monotherapy arm not applicable for this outcome measure
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Trametinib) | Treatment (Trametinib, Akt Inhibitor GSK2141795)
Number analyzed (Participants) | 0 | 11
Participants | 0 | 2

5. Secondary Outcome: Incidence of Adverse Event Reactions Reported According to CTCAE v4.0
Description: Reported by type, frequency, and severity.
Time Frame: From time of treatment start until treatment completion, an average of 1 year
Measure: Number; unit: Adverse Events
Arm/Group | Treatment (Trametinib) | Treatment (Trametinib, Akt Inhibitor GSK2141795)
Number analyzed (Participants) | 25 | 12
Adverse Events | 2 | 4

6. Other Pre Specified Outcome: Pharmacodynamic Markers of Trametinib
Description: Analyses will be descriptively summarized.
Time Frame: Baseline, day 1 of course 2, progression
Population: Data for this measure was not analyzed
Arm/Group | Treatment (Trametinib, Akt Inhibitor GSK2141795)
Number analyzed (Participants) | 0

7. Other Pre Specified Outcome: Chromosomal Abnormalities as Determined by FISH
Description: Analyses will be descriptively summarized.
Time Frame: At baseline
Population: Data for this measure was not analyzed
Arm/Group | Treatment (Trametinib, Akt Inhibitor GSK2141795)
Number analyzed (Participants) | 0

8. Other Pre Specified Outcome: Tumor Mutational Profile by Next Generation Sequencing
Description: Analyses will be descriptively summarized.
Time Frame: At baseline
Population: Data for this measure was not analyzed
Arm/Group | Treatment (Trametinib, Akt Inhibitor GSK2141795)
Number analyzed (Participants) | 0

9. Other Pre Specified Outcome: Change in RAS-MEK-ERK Activation Determined by Phospho-flow Cytometry and RPPA (Reversal Phase Protein Arrays)
Description: Analyses will be descriptively summarized.
Time Frame: At baseline
Population: Data for this measure was not analyzed
Arm/Group | Treatment (Trametinib, Akt Inhibitor GSK2141795)
Number analyzed (Participants) | 0

10. Other Pre Specified Outcome: Detection of RAS and RAF Mutations Using cfDNA
Description: Ultra-deep sequencing will be performed on cfDNA to assess the feasibility of detecting mutations of NRAS, KRAS and BRAF from peripheral blood samples.
Time Frame: Baseline and every even cycle and at progression, an average of 9 cycles (9 months)
Population: 64 cfDNA specimens from 53 Myeloma patients including 13 patients from this trial that were included in this analysis
Measure: Number; unit: MUTATIONS
Groups:
- Detection of KRAS Mutations Using cfDNA: Ultra-deep sequencing will be performed on cfDNA to assess the feasibility of detecting mutations of KRAS from peripheral blood samples.
- Detection of NRAS Mutations Using cfDNA: Ultra-deep sequencing will be performed on cfDNA to assess the feasibility of detecting mutations of NRAS from peripheral blood samples.
- Detection of BRAF Mutations Using cfDNA: Ultra-deep sequencing will be performed on cfDNA to assess the feasibility of detecting mutations of BRAF from peripheral blood samples.
Arm/Group | Detection of KRAS Mutations Using cfDNA | Detection of NRAS Mutations Using cfDNA | Detection of BRAF Mutations Using cfDNA
Number analyzed (Participants) | 22 | 13 | 7
MUTATIONS | 10 | 2 | 2

ADVERSE EVENTS:
Time Frame: From treatment start until 4 weeks after treatment end or death (whichever occurs first), for each patient, an average of 1 year.
Description: Adverse events collected as per protocol using CTCAE version 4.0
Arm/Group | Treatment (Trametinib, Akt Inhibitor GSK2141795)
All-Cause Mortality (participants affected / at risk) | 7/25
Serious Adverse Events (participants affected / at risk) | 15/25
Other Adverse Events (participants affected / at risk) | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Trametinib, Akt Inhibitor GSK2141795) (N=25)
Sepsis (Infections and infestations) | 6 — Sepsis
Lung infection (Infections and infestations) | 2 — Lung infection
Intracranial hemorrhage (Nervous system disorders) | 2 — Intracranial hemorrhage
NEOPLASMS BENIGN, MALIGNANT AND UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 — NEOPLASMS BENIGN, MALIGNANT AND UNSPECIFIED (INCL CYSTS AND POLYPS)-OTHER, PROGRESSIVE DISEASE
Confusion (Psychiatric disorders) | 3 — Confusion
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Trametinib, Akt Inhibitor GSK2141795) (N=25)
thrombocytopenia (Investigations) | 13 — Platelet count decreased
Nausea (Gastrointestinal disorders) | 14 — Nausea
Rash (Skin and subcutaneous tissue disorders) | 17 — Rash

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-23): https://cdn.clinicaltrials.gov/large-docs/98/NCT01989598/Prot_SAP_000.pdf